CLINICAL TRIAL: NCT01867801
Title: Portuguese Registry on Interventional Cardiology
Acronym: PRIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Portuguese Society of Cardiology (Other)
Collaborators: Portuguese Association of Interventional Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: RNCI
Record Dates: First submitted 2013-04-24; First posted 2013-06-04 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Coronary disease; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this Registry is creating a database management that allows continuous monitoring characteristics, evolution, prognostic indicators and management of patients undergoing coronary angioplasty in Portuguese Hospitals, and identify the appropriateness of clinical and interventional practice recommendations for diagnosis and treatment of coronary disease and monitoring its evolution.

DETAILED DESCRIPTION:
Cardiovascular disease remains the main cause of death in Portugal and approximately one quarter of these are directly to ischemic heart disease. In order to better characterize percutaneous coronary intervention in Portugal, the Portuguese Society of Cardiology has promoted the Portuguese registry on percutaneous coronary intervention.

This will include all adult patients (≥ 18 years), eligible for percutaneous coronary intervention (PCI) in accordance with PCI state-of-art recommendations (including unstable and stable coronary disease). The Cardiology department where the patient has been hospitalized is responsible for the patient inclusion in the study.

Excluded patients are those in whom the preferred treatment is Coronary Artery Bypass Graft (CABG), age under 18 years or life expectancy of less than 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with:

   * stable angina or,
   * stabilized angina pectoris or,
   * atypical chest pain or,
   * no chest pain but with documented silent ischemia
2. At least one stenosis is present of at least 50% in one major native epicardial coronary artery and supplying viable myocardium
3. Eligible for PCI
4. Informed consent

Exclusion Criteria:

1. Patients in whom the preferred treatment is CABG;
2. Contra-indication to dual antiplatelet therapy
3. Coronary artery disease precluding PCI
4. A life expectancy of less than 1 year
5. Age under 21

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to Portuguese hospitals for percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2002-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event rate (MACE) MACE: A composite of all cause death, documented Myocardial Infarction (MI), unplanned hospitalization leading to urgent revascularization. | 24 months

SECONDARY OUTCOMES:
Total mortality | 12 month
  Total mortality at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Marco Costa, MD, Principal Investigator — Portuguese Society of Cardiology
Locations (1):
- CNCDC, Coimbra, Portugal

REFERENCES:
- See also: Portuguese Society of Cardiology — http://www.spc.pt/spc